CLINICAL TRIAL: NCT01708603
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Induction and Maintenance Regimens of Brodalumab Compared With Placebo and Ustekinumab in Subjects With Moderate to Severe Plaque Psoriasis: AMAGINE-2
Brief Title: P3 Study Brodalumab in Treatment of Moderate to Severe Plaque Psoriasis
Acronym: AMAGINE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120103
Record Dates: First submitted 2012-09-12; First posted 2012-10-17 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: psoriasis, brodalumab, AMG 827
MeSH Terms: conditions — Psoriasis | interventions — brodalumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 210 mg brodalumab (Experimental): Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to schedule 1, 2, 3, or 4.
  Interventions: Drug: 210 mg brodalumab
- 140 mg brodalumab (Experimental): Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to schedule 1, 2, 3, or 4.
  Interventions: Drug: 140 mg brodalumab
- ustekinumab (Active Comparator): Administered by subcutaneous (SC) injection per the labeled dosing regimen.
  Interventions: Drug: ustekinumab
- Placebo (Placebo Comparator): Administered by subcutaneous (SC) injection until week 12. At week 12 participants are assigned to 210 mg brodalumab.
  Interventions: Drug: 210 mg brodalumab; Drug: placebo

INTERVENTIONS:
Drug: 210 mg brodalumab — 210 mg brodalumab administered SC
  Arms: 210 mg brodalumab; Placebo
Drug: 140 mg brodalumab — 140 mg brodalumab administered SC
  Arms: 140 mg brodalumab
Drug: ustekinumab — 45 mg or 90 mg ustekinumab administered SC per the labeled dosing regimen.
  Arms: ustekinumab
Drug: placebo — Placebo administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of brodalumab at two different doses

DETAILED DESCRIPTION:
.The purpose of this study is to assess the safety and efficacy of brodalumab at two different doses compared with placebo in participants with moderate to severe plaque psoriasis. A second purpose of this study is to assess the safety and efficacy brodalumab at two different doses compared with ustekinumab in participants with moderate to severe plaque psoriasis. A third purpose of this study is to assess the safety and efficacy of 4 maintenance regimens of brodalumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* Subject has involved body surface area (BSA) ≥ 10%, PASI ≥ 12, and sPGA ≥ 3 at screening and at baseline

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at (eg, eczema) that would interfere with study evaluations
* Subject has known history of Crohn's disease
* Subject has any other significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol
* Subject has not stopped using certain psoriasis therapies as defined in the study protocol
* Subject has previously used ustekinumab or any anti-IL-17 biologic therapy
* Subject is pregnant or breastfeeding, or planning to become pregnant while enrolled in the study
* Female subject is unwilling to use highly effective methods of birth control unless 2 years post-menopausal or surgically sterile

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1831 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (130):
- United States (59):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Vista, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Carmel, Indiana
  - Research Site, Plainfield, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Rockville, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, North Andover, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Fridley, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Gahanna, Ohio
  - Research Site, South Euclid, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
- Australia (8):
  - Research Site, Phillip, Australian Capital Territory
  - Research Site, Kogarah, New South Wales
  - Research Site, Benowa, Queensland
  - Research Site, Gold Coast, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Box Hill, Victoria
  - Research Site, Carlton, Victoria
  - Research Site, Parkville, Victoria
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Canada (13):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Jihlava
  - Research Site, Nový Jičín
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- France (10):
  - Research Site, Amiens
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Rouen
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Veszprém
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Poland (8):
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (10):
  - Research Site, Córdoba, AndalucÃ-a
  - Research Site, Seville, AndalucÃ-a
  - Research Site, Alcañiz, AragÃ³n
  - Research Site, Manacor, Balearic Islands
  - Research Site, Badalona, CataluÃ±a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, A Coruña, Galicia
  - Research Site, Alcorcón, Madrid
  - Research Site, Valencia, Valencia
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lebwohl MG, Armstrong AW, Alexis AF, Lain EL, Jacobson AA. Efficacy of Brodalumab in Patients with Psoriasis and Risk Factors for Treatment Failure: A Review of Post Hoc Analyses. Dermatol Ther (Heidelb). 2024 Oct;14(10):2709-2726. doi: 10.1007/s13555-024-01264-3. Epub 2024 Sep 12. PMID 39264399
- [Derived] Kokolakis G, Vadstrup K, Hansen JB, Carrascosa JM. Increased Skin Clearance and Quality of Life Improvement with Brodalumab Compared with Ustekinumab in Psoriasis Patients with Aggravating Lifestyle Factors. Dermatol Ther (Heidelb). 2021 Dec;11(6):2027-2042. doi: 10.1007/s13555-021-00618-5. Epub 2021 Oct 2. PMID 34606048
- [Derived] Gottlieb A, Lebwohl M, Liu C, Israel RJ, Jacobson A. Malignancy Rates in Brodalumab Clinical Studies for Psoriasis. Am J Clin Dermatol. 2020 Jun;21(3):421-430. doi: 10.1007/s40257-020-00512-4. PMID 32207067
- [Derived] McMichael A, Desai SR, Qureshi A, Rastogi S, Alexis AF. Efficacy and Safety of Brodalumab in Patients with Moderate-to-Severe Plaque Psoriasis and Skin of Color: Results from the Pooled AMAGINE-2/-3 Randomized Trials. Am J Clin Dermatol. 2019 Apr;20(2):267-276. doi: 10.1007/s40257-018-0408-z. PMID 30471012
- [Derived] Langley RG, Armstrong AW, Lebwohl MG, Blauvelt A, Hsu S, Tyring S, Rastogi S, Pillai R, Israel R. Efficacy and safety of brodalumab in patients with psoriasis who had inadequate responses to ustekinumab: subgroup analysis of two randomized phase III trials. Br J Dermatol. 2019 Feb;180(2):306-314. doi: 10.1111/bjd.17318. Epub 2018 Dec 27. PMID 30328108
- [Derived] Lebwohl M, Strober B, Menter A, Gordon K, Weglowska J, Puig L, Papp K, Spelman L, Toth D, Kerdel F, Armstrong AW, Stingl G, Kimball AB, Bachelez H, Wu JJ, Crowley J, Langley RG, Blicharski T, Paul C, Lacour JP, Tyring S, Kircik L, Chimenti S, Callis Duffin K, Bagel J, Koo J, Aras G, Li J, Song W, Milmont CE, Shi Y, Erondu N, Klekotka P, Kotzin B, Nirula A. Phase 3 Studies Comparing Brodalumab with Ustekinumab in Psoriasis. N Engl J Med. 2015 Oct;373(14):1318-28. doi: 10.1056/NEJMoa1503824. PMID 26422722
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Ustekinumab | Placebo
Started | 612 | 610 | 300 | 309
Completed | 597 | 588 | 291 | 300
Not Completed | 15 | 22 | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Ustekinumab | Placebo | Total
Number analyzed (Participants) | 612 | 610 | 300 | 309 | 1831
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.7) | 44.8 (12.8) | 45.4 (13.0) | 43.7 (12.9) | 44.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 197 | 95 | 90 | 573
  Male | 421 | 413 | 205 | 219 | 1258
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 2 | 8
  Asian | 19 | 25 | 12 | 12 | 68
  Native Hawaiian or Other Pacific Islander | 5 | 4 | 0 | 0 | 9
  Black or African American | 19 | 13 | 7 | 14 | 53
  White | 551 | 557 | 271 | 273 | 1652
  More than one race | 5 | 1 | 3 | 1 | 10
  Unknown or Not Reported | 10 | 8 | 6 | 7 | 31
Region of Enrollment [Number; unit: participants]
  Canada | 64 | 66 | 32 | 33 | 195
  Czechia | 18 | 20 | 7 | 8 | 53
  Netherlands | 5 | 6 | 3 | 3 | 17
  Austria | 6 | 8 | 2 | 4 | 20
  Hungary | 18 | 15 | 8 | 10 | 50
  United States | 286 | 281 | 140 | 144 | 851
  Poland | 130 | 132 | 65 | 64 | 391
  Australia | 40 | 39 | 20 | 19 | 118
  France | 14 | 13 | 9 | 8 | 44
  Portugal | 12 | 10 | 4 | 6 | 32
  Spain | 19 | 20 | 10 | 10 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Static Physician Global Assessment (sPGA) Score Success (Score of 0 or 1) at Week 12
Description: Measures the physician's impression of the disease at a single point, and a dynamic form in which the physician assesses the global improvement from baseline. Success is defined by a score of 0 or 1 (clear to almost clear).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Ustekinumab: Administered by subcutaneous (SC) injection until week 12. Participants using Ustekinumab were not rerandomized at week 12, and continued to receive ustekinumab.
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Ustekinumab
Number analyzed (Participants) | 612 | 610 | 309 | 300
Participants | 481 | 354 | 12 | 183

2. Primary Outcome: Percentage of Participants With Psoriasis Area Severity Index (PASI) 75 at Week 12
Description: to evaluate the efficacy of Brodalumab (210mg every 2 weeks, and 140mg every 2 weeks) in subjects with moderate to severe plaque psoriasis, as measured by the proportion of subjects achieving 75% improvement in Psoriasis Area and Severity Index, PASI75 at week 12.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Brodalumab Placebo
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Ustekinumab
Number analyzed (Participants) | 612 | 610 | 309 | 300
Participants | 528 | 406 | 25 | 210

3. Primary Outcome: Percentage of Participants With Psoriasis Area Severity Index (PASI) 100 at Week 12
Description: to evaluate the efficacy of Brodalumab (210mg Q2W) in clearing psoriasis as measured by the proportion of subjects achieving PASI 100 at week 12.
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Brodalumab 210mg: Brodalumab 210mg Q2W
- Brodalumab 140mg: Brodalumab 140mg Q2W
- Ustekinumab: Ustekinumab administered in a dose of 45mg in a prefilled syringe of 0.5mL
Arm/Group | Brodalumab 210mg | Brodalumab 140mg | Placebo | Ustekinumab
Number analyzed (Participants) | 612 | 610 | 309 | 300
Participants | 272 | 157 | 2 | 65

ADVERSE EVENTS:
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Ustekinumab | Placebo
Serious Adverse Events (participants affected / at risk) | 6/612 | 13/610 | 4/300 | 8/309
Other Adverse Events (participants affected / at risk) | 354/612 | 365/610 | 177/300 | 165/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=612) | 140 mg Brodalumab (N=610) | Ustekinumab (N=300) | Placebo (N=309)
Pancreatitis Acute (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Blood Glucose Increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Diabetes Mellitus Inadequate Control (General disorders) | 0 | 0 | 0 | 1
Dysponea (General disorders) | 0 | 0 | 0 | 1
Escherichia Urinary tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Noncardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1
Syncope (General disorders) | 0 | 0 | 0 | 1
Alcohol Abuse (General disorders) | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Anteriosclerosis (Cardiac disorders) | 0 | 1 | 0 | 0
Carbon Monoxide Poisining (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cerbebral Infarction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Chondromalacia (General disorders) | 0 | 1 | 0 | 0
Chondropathy (General disorders) | 0 | 1 | 0 | 0
Drug Detoxification (General disorders) | 0 | 1 | 0 | 0
Fibromyalgia (General disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Joint Capsule Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Vertigo (General disorders) | 0 | 0 | 1 | 0
Acute Coronary Syndrome (Vascular disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=612) | 140 mg Brodalumab (N=610) | Ustekinumab (N=300) | Placebo (N=309)
Nasopharyngitis (Infections and infestations) | 45 | 45 | 18 | 14
Upper respiratory Tract infection (Infections and infestations) | 33 | 30 | 20 | 23
Bronchitis (Infections and infestations) | 12 | 3 | 4 | 3
Sinusitis (Infections and infestations) | 7 | 3 | 7 | 3
Urinary tract Infection (Infections and infestations) | 3 | 8 | 2 | 4
Influenza (Infections and infestations) | 7 | 7 | 1 | 1
Viral Upper respiratory Tract Infection (Infections and infestations) | 6 | 5 | 3 | 0
Gastroenteritis (Infections and infestations) | 3 | 3 | 2 | 4
Rhinitis (Infections and infestations) | 2 | 3 | 4 | 2
Pharyngitis (Infections and infestations) | 7 | 3 | 1 | 0
Folliculitis (Infections and infestations) | 7 | 3 | 1 | 0
Oral Herpes (Infections and infestations) | 2 | 2 | 4 | 0
Conjuncitvitus (Infections and infestations) | 2 | 3 | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 5 | 0 | 1
Laryngitis (Infections and infestations) | 3 | 2 | 0 | 1
Tooth Infection (Infections and infestations) | 2 | 1 | 2 | 1
Otitis Media (Infections and infestations) | 4 | 1 | 1 | 0
Skin Infection (Infections and infestations) | 2 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 33 | 9 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 17 | 4 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 10 | 9 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 4 | 11 | 0 | 1
Muskuloskelital Pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 13 | 2 | 4
Nausea (Gastrointestinal disorders) | 11 | 9 | 5 | 5
Toothache (Gastrointestinal disorders) | 7 | 6 | 6 | 4
Abdominal Pain (Gastrointestinal disorders) | 4 | 8 | 1 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 10 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 5 | 3 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4 | 3 | 1
Dry Mouth (Gastrointestinal disorders) | 2 | 5 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 19 | 6 | 7
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 3
Acne (Skin and subcutaneous tissue disorders) | 6 | 3 | 2 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 5 | 1 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 0
headache (Nervous system disorders) | 31 | 35 | 12 | 9
Paraesthesia (Nervous system disorders) | 3 | 4 | 2 | 1
Sciatica (Nervous system disorders) | 3 | 5 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 2
Migrane (Nervous system disorders) | 2 | 1 | 2 | 0
Sinus headache (Nervous system disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 16 | 11 | 12 | 2
Pyrexia (General disorders) | 8 | 6 | 2 | 0
Peripheral Swelling (General disorders) | 4 | 4 | 0 | 3
Asthenia (General disorders) | 5 | 6 | 4 | 1
Odema Peripheral (General disorders) | 2 | 2 | 1 | 4
Injection Site Pain (General disorders) | 3 | 5 | 0 | 1
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 13 | 9 | 3 | 5
Laceration (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 3
Joint Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 1 | 6
Hyperuricaemia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 4
Gout (Metabolism and nutrition disorders) | 3 | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days